CLINICAL TRIAL: NCT05004896
Title: Repeated Ketamine Infusions for Treatment-Resistant Bipolar Disorder: A Randomized, Double-blind, Midazolam-controlled, Phase II Clinical Trial
Brief Title: Ketamine for Treatment-Resistant Bipolar Disorder
Acronym: KET-BD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joshua Rosenblat (Other)
Responsible Party: Sponsor-Investigator, Joshua Rosenblat, Principal Investigator, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-5560
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Four infusions of ketamine will be administered over two weeks. The first two infusions will be dosed at 0.5mg/kg over a period of 40 minutes. For infusions 3 and 4, patients will be flexibly dosed between 0.5 mg/kg to 0.75 mg/kg, depending on clinical response to first two infusions.
  Interventions: Drug: Ketamine Hydrochloride
- Midazolam (Active Comparator): Four infusions of midazolam will be administered over two weeks. The first two infusions will be dosed at 0.02mg/kg over a period of 40 minutes. For infusions 3 and 4, patients will be flexibly dosed between 0.02 mg/kg to 0.03 mg/kg, depending on clinical response to first two infusions.
  Interventions: Drug: Midazolam Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — 36 patients will receive ketamine hydrochloride, over four infusions, flexibly dosed between 0.5 mg/kg to 0.75 mg/kg
  Arms: Ketamine
Drug: Midazolam Hydrochloride — 36 patients will receive midazolam hydrochloride, over four infusions, flexibly dosed between 0.02 mg/kg to 0.03 mg/kg
  Arms: Midazolam

SUMMARY:
Growing evidence has supported rapid and robust antidepressant effects with subanesthetic doses of intravenous (IV) ketamine for treatment resistant depression (TRD). However, no completed or ongoing randomized control trials (RCTs) have evaluated the effects of repeated doses of IV ketamine for a homogenous sample of patients with treatment-resistant bipolar disorder (TRBD). The primary research goal is to determine the acute antidepressant efficacy, safety and tolerability of four repeated sub-anesthetic doses of IV ketamine in moderate to severe TRBD. Secondary aims include evaluating effects of IV ketamine on suicidal ideations, quality of life, function and duration of effects. Herein, a two-site (University Health Network and Ontario Shores Centre for Mental Health Sciences), phase II, double-blinded, midazolam-controlled, two-week RCT evaluating the efficacy, safety and tolerability of four flexibly-dosed adjunctive ketamine infusions (0.5-0.75mg/kg infused over 40 minutes) for acute treatment of moderate to severe TRBD (type I & II) is proposed. The primary outcome will be Montgomery-Åsberg Depression Rating Scale (MADRS) scores, determining the between group difference in change from baseline to day 14, using analysis of covariance (ANCOVA), with 14-day MADRS as the outcome and baseline MADRS and stratification variables (sex, bipolar type) as covariates. Secondary outcomes include evaluating response and remission rates, safety, tolerability (including treatment-emergent mania), and effects on suicidality, anxiety, quality of life, function and the duration of effects (to day 28).

ELIGIBILITY:
Inclusion Criteria

1. Provide written, voluntary informed consent prior to study enrollment. Substitute decision makers will not be allowed to consent to study on a potential patient's behalf.
2. Male or female between the age of 21 to 65, inclusive.
3. Meets DSM-5 criteria for Bipolar I or II Disorder, currently experiencing a Major Depressive Episode without psychotic features. Diagnosis will be confirmed using the Mini-International Neuropsychiatric Interview (MINI) conducted by a delegated physician or trained research study while assessing eligibility.
4. Patient must present with a moderate to severe depressive episode, as determined by the MADRS score greater than 21.
5. Current depressive episode has inadequate response to two or more adequate first-line treatment trials for bipolar depression, as per the 2018 CANMAT Bipolar Disorder Guidelines. First line treatment trials include the use of lithium, valproate, carbamazepine, lamotrigine and/or any antipsychotic medication.
6. Patient must be receiving guideline-concordant pharmacotherapy without changes in the last month, including a therapeutic dose of a guideline-concordant mood stabilizer/antipsychotic.

Exclusion Criteria

1. Currently exhibiting symptoms of mania, hypomania, or mixed state bipolar, as determined by the Young Mania Rating Scale (YMRS) score greater than 12.
2. Current symptoms of psychosis or a substance use disorder within the past 3 months. History of psychotic features during a mood episode will not be excluded.
3. History of neurological disorders (including, but not limited to, uncontrolled seizure disorder, history of stroke within past 12 months, major head injuries, aneurysmal vascular disease [including thoracic and abdominal aorta, intracranial, and peripheral arterial vessels], arteriovenous malformation, or intracerebral hemorrhage)
4. Lifetime history of a primary psychotic disorder (including, but not limited to, schizophrenia or schizoaffective disorder)
5. Lifetime history of ketamine use disorder
6. Presence of active suicidality, requiring involuntary inpatient treatment or recent suicide attempts within the past 3 months.
7. Presence of a contraindication to ketamine or midazolam, including a drug allergy, uncontrolled hypertension (baseline systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg), low or labile blood pressure, myocardial infarction within past 12 months, cardiac arrhythmia, moderate to severe hepatic impairment (i.e., Child-Pugh score of B or C), moderate or severe renal impairment (glomerular filtration rate (GFR) < 45 milliliters/min) , heart failure, or coronary artery disease
8. Pregnant or breastfeeding women or women who intend to get pregnant. Patients who are sexually active must agree to use a highly effective contraceptive method (as outlined in section 5.11).
9. Use of prohibited concomitant medications, including other forms of ketamine or esketamine, benzodiazepines, stimulants, alcohol, and medical or recreational cannabis taken during the trial at a specific prohibited time.
10. Use of ketamine in the 30 days leading up to the patient's entry in the trial.
11. Use of monoamine oxidase inhibitors (MAOIs) at least two weeks prior to receiving study treatment.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Change in depression severity using the Montgomery Asberg Depression Rating Scale (MADRS) | 4 weeks
  The MADRS is a clinician-rated scale measuring depression severity. It consists of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60. A higher score is indicative of greater depressive severity. Response rates are defined as > 50% decrease and Remission < 12 actual score.

SECONDARY OUTCOMES:
Recruitment and Retention Rate | 4 weeks
  The feasibility of ketamine as a treatment in bipolar disorder will be measured by recruitment and retention rates.
Treatment-Emergent Adverse Events | 4 weeks
  Treatment-emergent adverse events will be assessed using patient-reported adverse events.
Suicidality | 4 weeks
  Suicidality will be assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS) which is a clinical assessment used to assess suicidal ideation and suicidal behaviour. It measures the incidence of suicidality via "yes" or "no" questions as well as the severity of suicidal ideation if present on a scale of 1 to 5 with 5 being the most severe.
Treatment-Emergent Mania | 4 weeks
  Treatment-emergent mania will be assessed using the Young Mania Rating Scale (YMRS) which is a clinical assessment used to evaluate manic symptoms and their severity. It consists of 11 items with a maximum possible score of 60, with higher scores indicating more severe manic symptoms.
Quality of Life (QOL) | 4 weeks
  Quality of life will be assessed using the Quality of Life-BD (QOL.BD) scale, which contains 56 questions over 12 domains. It uses a 5-component scale that evaluates mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This scale is numbered from 56 to 280, 280 indicating a high quality of life, while 56 denotes a low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rosenblat, MD, MSc, Principal Investigator — Toronto Western Hospital, Psychiatry
Locations (3):
- Canada (3):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: No